CLINICAL TRIAL: NCT02639377
Title: Efficacy of 0.12% Chlorhexidine Gluconate for Peri-implant Mucositis and Gingivitis: a Randomised Controlled Clinical Trial
Brief Title: Efficacy of 0.12% Chlorhexidine Gluconate for Peri-implant Mucositis and Gingivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Karyna de Melo Menezes, Principal Investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFRN-2
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Mucositis; Gingivitis
Keywords: Dental Implantation; Chlorhexidine gluconate
MeSH Terms: conditions — Mucositis; Gingivitis | interventions — chlorhexidine gluconate; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine gluconate (Experimental): 15 ml of solution every 12 hours, twice a day, 30 minutes after brushing, for 14 days
  Interventions: Drug: Chlorhexidine gluconate
- Placebo (Placebo Comparator): 15 ml of solution every 12 hours, twice a day, 30 minutes after brushing, for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chlorhexidine gluconate
  Other Names: Chlorhexidine
  Arms: Chlorhexidine gluconate
Drug: Placebo — Solution chemical manufactured to mimic 0.12% chlorhexidine mouthwash
  Other Names: placebo solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to analyze the efficacy of 0.12% chlorhexidine gluconate as a chemical adjuvant for the treatment of peri-implant mucositis in single implants compared with homologous teeth with gingivitis, in a non-surgical treatment protocol with a six-month follow-up.

DETAILED DESCRIPTION:
The following clinical parameters were evaluated in both test and control groups; visible plaque index (VPI) and gingival bleeding index (GBI) were obtained for full mouth (IPV and ISG) and for each implant and teeth (VPI implant; VPI teeth; GBI implant; GBI teeth). For statistical purposes, percentages of faces with biofilm and marginal bleeding at teeth and implants were calculated. These parameters were evaluated at baseline and at one, three and six months post-therapy.

Probing depth (PD implant; PD teeth) and bleeding on probing (BOP implant; BOP teeth) were collected for all implants and teeth with a North Carolina periodontal probe at six sites. After data collection, an arithmetic averages of the sites with bleeding on probing and probing depths were calculated at baseline, three and six months. The peri-implant and periodontal biotype for each implant and teeth was rated as thin or thick, according to probe transparency during probing depth.

ELIGIBILITY:
Inclusion Criteria:

* Systemically-healthy partially edentulous patients rehabilitated with functional dental implants and prostheses for at least 1 year;
* Patients had been diagnosed with peri-implant mucositis, probing depth up to 5 mm, bleeding on probing and no radiographic evidence of bone loss beyond the first two threads of the implant;
* Patients had been diagnosed with gingivitis in homologous teeth to implants.

Exclusion Criteria:

* Non-smokers and not in maintenance therapy;
* Periodontal treatment during the last six months;
* Have not used antimicrobial (systemic or topical), anti-inflammatory or immunosuppressive drugs during the six months preceding the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing | baseline
Bleeding on probing | three months
Bleeding on probing | six months

SECONDARY OUTCOMES:
Probing depth | baseline and at three and six months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno CV Gurgel, Doctor, Study Director — Universidade Federal do Rio Grande do Norte

IPD SHARING:
Plan to Share IPD: No